CLINICAL TRIAL: NCT05383820
Title: Effect of Paracetamol and Ketorolac on RANK-L Levels in Patients Starting Orthodontic Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Juan Ramon Gomez Sandoval, principal investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CI04820
Record Dates: First submitted 2021-09-04; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Malocclusion; Pain, Acute
Keywords: Orthodontics; RANK-L; Ketorolac; Paracetamol; Gingival crevicular fluid
MeSH Terms: conditions — Malocclusion; Acute Pain | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: A double-blind clinical trial will be carried out with a placebo control group and random drug allocation. Patients who begin orthodontic treatment in the Orthodontic Specialty of the Comprehensive Dental Clinics of the University Center for Health Sciences and who decide to participate in the study with the signing of informed consent will be included. Three groups will be formed with 8 patients in each one.
  The first group will be administered with Placebo (calcined magnesia), the second group with Ketorolac and the third group with Paracetamol, for all groups the medication will be one capsule every 6 hours for 5 days all study subjects will be sampled Gingival Crevicular Fluid (LGC), Visual Analogue Pain Scale (APS) and Intermolar Space (IS).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded, the orthodontist performing the clinical intervention and the investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo (calcined magnesia) in capsules, one capsule every 8 hours for 5 days.
  Interventions: Drug: Ketorolac
- Ketorolac (Experimental): Ketorolac 10 mg capsules, one capsule every 8 hours (30 mg daily) for 5 days.
  Interventions: Drug: Ketorolac
- Paracetamol (Active Comparator): Paracetamol capsules of 500 mg, one capsule every 8 hours (1.5 g per day) for 5 days.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — The first group will be administered with Placebo (calcined magnesia), the second group with Ketorolac and the third group with Paracetamol, for all groups the medication will be one capsule every 6 hours for 5 days all study subjects will be sampled Gingival Crevicular Fluid (LGC), Visual Analogue Pain Scale (APS) and Intermolar Space (IS).
  Other Names: Parcetamol

SUMMARY:
Due to the high prevalence of malocclusions in Mexico and the existing concern to improve aesthetics, function (chewing), or both, patients resort to orthodontic treatment. The patient may experience pain during treatment due to the release of different chemical mediators such as RANK-L. Analgesic and anti-inflammatory medications such as acetaminophen and ketorolac are used to control pain during orthodontic tooth movement. These drugs can inhibit the expression of RANK-L which can affect tooth movement, inhibiting bone remodeling. The orthodontist should indicate the drug that is safest for the patient without affecting treatment or tooth movement.

DETAILED DESCRIPTION:
Objective: To evaluate the association of RANK-L levels with the administration of paracetamol and ketorolac in patients starting orthodontic treatment.

Material and methods: A double-blind clinical trial will be carried out with a placebo control group and random drug allocation. Patients who begin orthodontic treatment in the Orthodontic Specialty of the Comprehensive Dental Clinics of the University Center for Health Sciences and who decide to participate in the study with the signing of informed consent will be included. Three groups will be formed with 8 patients in each one.

The first group will be administered with Placebo (calcined magnesia), the second group with Ketorolac and the third group with Paracetamol, for all groups the medication will be one capsule every 6 hours for 5 days all study subjects will be sampled Gingival Crevicular Fluid (LGC), Visual Analogue Pain Scale (APS) and Intermolar Space (IS).

Measurements will be made four times; baseline, 24 h, 48 h, and on day 5 of initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between 18 and 27 years of age
* Periodontally and systematically healthy
* Attended the Orthodontic Clinic of the University of Guadalajara
* Who required the use of dental spacers in at least one quadrant were included

Exclusion Criteria:

* Patients who have previously had orthodontic treatment or are under orthodontic treatment
* Who have an allergy to ketorolac or paracetamol
* Who are under pharmacological treatment and/or using contraceptives
* Pregnant or lactating women, as well as those who consume alcohol were not included or tobacco.

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-12-18 (Estimated)

PRIMARY OUTCOMES:
Leves RANK-L | Baseline, 24 hours, 48 hours, and on day 5 of initiation of treatment.
  Leves Gingival Crevicular Fluid of RANK-L

SECONDARY OUTCOMES:
Pain scale | Baseline, 24 hours, 48 hours, and on day 5 of initiation of treatment.
  Visual Analogue Pain Scale (APS)
Intermolar Space (IS) | 5 days of initiation of treatment.
  It is the space between the molars

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Ramón Gómez Sandoval, Guadalajara, Jaisco, Mexico

IPD SHARING:
Plan to Share IPD: No